CLINICAL TRIAL: NCT02861586
Title: Double Blinded, Randomized, Priorix®- and Placebo-controlled, Trial to Evaluate the Optimal Dose of MV-CHIK Vaccine (Against Chikungunya Virus) in Regard to Immunogenicity, Safety and Tolerability in Healthy Volunteers
Brief Title: Phase II Study to Evaluate Safety and Immunogenicity of a Chikungunya Vaccine
Acronym: MV-CHIK-202
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Themis Bioscience GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MV-CHIK-202; 2015-004037-26 (EudraCT Number); V184-002 (Other: Merck & Co., protocol ID since aquisition in May 2020)
Record Dates: First submitted 2016-07-28; First posted 2016-08-10 (Estimated); Results first posted 2021-06-08 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Chikungunya Virus Infection
Keywords: Chikungunya, infectious disease
MeSH Terms: conditions — Chikungunya Fever; Communicable Diseases | interventions — Measles-Mumps-Rubella Vaccine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Treatment Group A; MV-CHIK low (Experimental): 60 subjects will receive i.m. vaccinations with MV-CHIK low dose (5xE4 (± 0.5 log) TCID50 per 0.3 mL) on study day 0 and 28, placebo on day 196.
  Physical examinations, vital signs, pregnancy tests for females, inquiry of adverse events and collection of immunogenicity blood samples will be performed during all visits.
  Interventions: Biological: MV-CHIK low dose; Biological: physiological saline solution
- Treatment Group A/C; Priorix® (Active Comparator): 20 subjects will receive i.m. vaccinations with Priorix® on study day 0 and 28, placebo on day 196.
  Physical examinations, vital signs, pregnancy tests for females, inquiry of adverse events and collection of immunogenicity blood samples will be performed during all visits.
  Interventions: Biological: Priorix®; Biological: physiological saline solution
- Treatment Group B; MV-CHIK low (Experimental): 60 subjects will receive i.m. vaccinations with placebo on study day 0. MV-CHIK low dose (5xE4 (± 0.5 log) TCID50 per 0.3 mL) on day 28 and MV-CHIK boosting dose on day 196.
  Physical examinations, vital signs, pregnancy tests for females, inquiry of adverse events and collection of immunogenicity blood samples will be performed during all visits.
  Interventions: Biological: MV-CHIK low dose; Biological: physiological saline solution
- Treatment Group B/D; Priorix® (Active Comparator): 20 subjects will receive i.m. vaccinations with placebo on study day 0, Priorix® on day 28 and one boosting dose with Priorix® on day 196.
  Physical examinations, vital signs, pregnancy tests for females, inquiry of adverse events and collection of immunogenicity blood samples will be performed during all visits.
  Interventions: Biological: Priorix®; Biological: physiological saline solution
- Treatment Group C; MV-CHIK high (Experimental): 60 subjects will receive i.m. vaccinations with MV-CHIK high dose (5xE5 (± 0.5 log) TCID50 per 0.3 mL) on study day 0 and 28, placebo on day 196.
  Physical examinations, vital signs, pregnancy tests for females, inquiry of adverse events and collection of immunogenicity blood samples will be performed during all visits.
  Interventions: Biological: MV-CHIK high dose; Biological: physiological saline solution
- Treatment Group D; MV-CHIK high (Experimental): 60 subjects will receive i.m. vaccinations with placebo on study day 0, MV-CHIK high dose (5xE5 (± 0.5 log) TCID50 per 0.3 mL) on study day 28 and MV-CHIK boosting dose on day 196.
  Physical examinations, vital signs, pregnancy tests for females, inquiry of adverse events and collection of immunogenicity blood samples will be performed during all visits.
  Interventions: Biological: MV-CHIK high dose; Biological: physiological saline solution
- Measles Booster Group 1 (Experimental): 20 subjects will receive i.m. vaccinations with Priorix® on study day -28, MV-CHIK on day 0 and 28 and placebo on day 168 and 196.
  Physical examinations, vital signs, pregnancy tests for females, inquiry of adverse events and collection of immunogenicity blood samples will be performed during all visits.
  Interventions: Biological: MV-CHIK low dose; Biological: Priorix®; Biological: physiological saline solution
- Measles Booster Group 2 (Experimental): 20 subjects will receive i.m. vaccinations with Priorix® on study day -28, placebo on day 0 and 28 and MV-CHIK on day 168 and 196.
  Physical examinations, vital signs, pregnancy tests for females, inquiry of adverse events and collection of immunogenicity blood samples will be performed during all visits.
  Interventions: Biological: MV-CHIK low dose; Biological: Priorix®; Biological: physiological saline solution

INTERVENTIONS:
Biological: MV-CHIK low dose — recombinant measles virus vaccine expressing Chikungunya virus antigens, powder for suspension for injection, 5xE4 (± 0.5 log) TCID50/dose
  Other Names: vaccine against Chikungunya
  Arms: Measles Booster Group 1; Measles Booster Group 2; Treatment Group A; MV-CHIK low; Treatment Group B; MV-CHIK low
Biological: MV-CHIK high dose — recombinant measles virus vaccine expressing Chikungunya virus antigens, powder for suspension for injection; 5xE5 (± 0.5 log) TCID50/dose
  Other Names: vaccine against Chikungunya
  Arms: Treatment Group C; MV-CHIK high; Treatment Group D; MV-CHIK high
Biological: Priorix® — lyophilized mixed preparation containing the attenuated Schwarz measles virus strain, the RIT 4385 strain of mumps virus (derived from the Jeryl Lynn strain) and the Wistar RA 27/3 rubella virus strain. Powder and solvent for suspension for injection
  Other Names: vaccine against Measles, Mumps and Rubella
  Arms: Measles Booster Group 1; Measles Booster Group 2; Treatment Group A/C; Priorix®; Treatment Group B/D; Priorix®
Biological: physiological saline solution — sterile physiological saline solution 0.9% used as placebo
  Other Names: 0.9% sodium chloride (NaCl)

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of a novel vaccine against Chikungunya virus after one or two vaccinations by comparison of two different dose levels.

DETAILED DESCRIPTION:
This is a double blinded, block-randomized, active- and placebo controlled, phase II trial, comparing two dose levels by assessing immunogenicity, safety and tolerability of MV-CHIK (a novel vaccine against Chikungunya virus).

Healthy male and female subjects aged 18-55 years will be randomized to one of six treatment groups (A, B, C. D, M1 or M2) differing in dosage and scheduling of vaccinations. Group A-D will be split in one arm receiving MV-CHIK and one control-arm receiving Priorix®.

All subjects of group A. B, C and D will receive three i.m. injections on study day 0, 28 and 196. Subjects of group A and B will receive MV-CHIK low dose or control-vaccine Priorix® (or equivalent measles vaccine) and subjects of group C and D will be treated with MV-CHIK high dose or control-vaccine (Priorix® or equivalent measles vaccine).

All subjects of group A, B, C and D additionally will be randomized to one of two treatment sequences: group A and C will receive MV-CHIK or control-vaccine Priorix® on study day 0 and 28, followed by placebo on day 196, and group B and D receive placebo on day 0 and MV-CHIK or Priorix® on day 28, followed by an additional vaccination of the same product on day196 (boosting vaccination).

All subjects of the measles booster group M1 and M2 will receive five i.m. injections on study day -28, 0, 28, 168 and 196. The first vaccination will be Priorix® (or equivalent measles vaccine) on study day -28. Group M1 will receive MV-CHIK vaccinations on day 0 and day 28 and placebo on day 168 and 196. Group M2 will receive placebo on day 0 and 28 and MV-CHIK on day 168 and on day 196.

All subjects will be followed for safety and immunogenicity evaluation until day 224. Study duration per subject is estimated to be 33-37 weeks (~8 months), respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent obtained before any trial-related activities.
2. Ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to cooperate with the investigator and to comply with the requirements of the entire study
3. Available for the duration of the trial
4. Healthy men or women aged >18 and <55 years
5. In female subjects either childbearing potential terminated by surgery or one year post-menopausal, or a negative urine pregnancy test during screening and the willingness not to become pregnant during the entire study period by practicing reliable methods of contraception as specified in protocol
6. Normal findings in medical history and physical examination or the investigator considers all abnormalities to be clinically irrelevant
7. Normal laboratory values or the investigator considers all abnormalities to be clinically irrelevant (unless otherwise specified in exclusion criteria)

Exclusion Criteria:

1. Participation in another clinical study within the past month in which the subject has been exposed to an investigational product (pharmaceutical product or placebo or device) or planned concurrent participation in another clinical study during the study period
2. History of immunodeficiency, known human immunodeficiency virus (HIV) infection, current hepatitis B/C infection,
3. Drug addiction including alcohol dependence
4. Inability or unwillingness to avoid more than the usual intake of alcohol during the 48 hours after vaccination (not more than 20g alcohol per day, which equals 0.5 L beer or 0.25 L of wine)
5. Persons who are accommodated in an institution on court or official order.
6. Persons in direct relationship with the sponsor, an Investigator or other study site staff. Direct relationship includes relatives or close dependents (children, spouse/partner, siblings or parents), as well as employees (site or sponsor).
7. Non-study licensed vaccines: vaccination within 4 weeks prior to first vaccination or planning to receive any non-study vaccine during the study period.
8. Measles vaccination or booster within the last 5 years or during the clinical study
9. Prior receipt of any Chikungunya vaccine
10. Blood donations during 1 month prior to Screening Visit and throughout the study
11. Recent infection (within 1 week prior to Screening Visit) (If non-serious, can be basis for temporary deferral)
12. Relevant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, hematological, endocrine, inflammatory or neurological diseases, that in the opinion of the investigator may interfere with the aim of the study
13. History of neoplastic disease (excluding non-melanoma skin cancer that was successfully treated) within the past 5 years or a history of any hematological malignancy.
14. History of autoimmune disease (e.g. rheumatoid arthritis, systemic lupus erythematosus (SLE), autoimmune thyroid disease).
15. History of moderate or severe arthritis or arthralgia within the past 3 months prior to Screening Visit.
16. Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the study protocol.
17. History of severe adverse reactions to vaccine administration, including anaphylaxis and related symptoms, such as urticaria, respiratory difficulty, angioedema and abdominal pain to vaccines, or history of allergic reaction likely to be exacerbated by any component of the vaccine.
18. History of anaphylaxis to drugs or major allergic reactions in general, which the investigator considers may compromise the safety of the volunteers
19. Clinically relevant abnormal laboratory values indicative of physical illness

    * Hematology: hemoglobin, hematocrit, erythrocyte count, differential white blood count, platelets
    * Chemistry: creatinine (≥1.7 mg/dL), potassium, sodium, calcium, aspartate transaminase/alanine aminotransferase (AST/ALT) ≥ 2.6 upper limit of normal (ULN), alkaline phosphatase, bilirubin
    * Coagulation parameter: prothrombin time (PT), activated partial thromboplastin time (aPTT), fibrinogen according to the evaluation of the principle investigator
    * Urinalysis according to the evaluation of the principle investigator
20. Use of medication during 2 weeks before the first vaccination and throughout the study, which the investigator considers may affect the validity of the study except hormonal contraception in female subjects; prior to taking any medication during 72 h prior to the first vaccination, the study center should be consulted.
21. Immunosuppressive drugs: use of corticosteroids (excluding topical preparations) or immunosuppressive drugs within 30 days prior to vaccination, or anticipated use during the trial.
22. Receipt of blood products or immunoglobulins within 120 days prior to Screening Visit or anticipated receipt of any blood products or immunoglobulin during the trial.
23. Pregnancy (positive pregnancy test at screening or during study phase), lactation or unreliable contraception in female subjects with child-bearing potential (for details please refer to section 8.3.6)
24. Subjects with any condition which in the opinion of the investigator makes the subject unsuitable for inclusion
25. Individuals who are living and/or working with severely immunocompromised people, children under 15 months old or pregnant women.
26. Inability or unwillingness to provide informed consent and to abide by the requirements of the study
27. Refusal to allow storage of specimens for future research.
28. Regular blood plasma donations

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 263 (Actual)
Dates: Start 2016-08-17 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2018-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (4):
- Austria (2):
  - Hansa Sanatorium GmbH, Graz
  - Medical University Vienna, Department of Clinical Pharmacology, Vienna
- Germany (2):
  - Berliner Center for Travel- and Tropical Medicine, Berlin
  - Medicinal University Rostock, Department for Tropical Medicin and infectious diseases, Rostock

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramsauer K, Schwameis M, Firbas C, Mullner M, Putnak RJ, Thomas SJ, Despres P, Tauber E, Jilma B, Tangy F. Immunogenicity, safety, and tolerability of a recombinant measles-virus-based chikungunya vaccine: a randomised, double-blind, placebo-controlled, active-comparator, first-in-man trial. Lancet Infect Dis. 2015 May;15(5):519-27. doi: 10.1016/S1473-3099(15)70043-5. Epub 2015 Mar 2. PMID 25739878
- [Derived] Tschismarov R, Zellweger RM, Koh MJ, Leong YS, Low JG, Ooi EE, Mandl CW, Ramsauer K, de Alwis R. Antibody effector analysis of prime versus prime-boost immunizations with a recombinant measles-vectored chikungunya virus vaccine. JCI Insight. 2021 Nov 8;6(21):e151095. doi: 10.1172/jci.insight.151095. PMID 34582377
- [Derived] Reisinger EC, Tschismarov R, Beubler E, Wiedermann U, Firbas C, Loebermann M, Pfeiffer A, Muellner M, Tauber E, Ramsauer K. Immunogenicity, safety, and tolerability of the measles-vectored chikungunya virus vaccine MV-CHIK: a double-blind, randomised, placebo-controlled and active-controlled phase 2 trial. Lancet. 2019 Dec 22;392(10165):2718-2727. doi: 10.1016/S0140-6736(18)32488-7. Epub 2018 Nov 5. PMID 30409443

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 322 participants screened for eligibility, 263 participants randomized
Pre-assignment Details: 59 screening failures (33 withdrawal of consent, 26 violation of in-/exclusion criteria)
Groups:
- Treatment Group A; MV-CHIK Low: Participants received i.m. vaccinations with MV-CHIK low dose (5xE4 (± 0.5 log) TCID50 per 0.3 mL) on study day 0 and 28, placebo on day 196. MV-CHIK low dose: recombinant measles virus vaccine expressing Chikungunya virus antigens, powder for suspension for injection, 5xE4 (± 0.5 log) TCID50/dose physiological saline solution: sterile physiological saline solution 0.9% used as placebo
- Treatment Group A/C; Priorix®: Participants received i.m. vaccinations with Priorix® on study day 0 and 28, placebo on day 196. Priorix®: lyophilized mixed preparation containing the attenuated Schwarz measles virus strain, the RIT 4385 strain of mumps virus (derived from the Jeryl Lynn strain) and the Wistar RA 27/3 rubella virus strain. Powder and solvent for suspension for injection physiological saline solution: sterile physiological saline solution 0.9% used as placebo
- Treatment Group B; MV-CHIK Low: Participants received i.m. vaccinations with placebo on study day 0, MV-CHIK low dose (5xE4 (± 0.5 log) TCID50 per 0.3 mL) on day 28 and MV-CHIK boosting dose on day 196. MV-CHIK low dose: recombinant measles virus vaccine expressing Chikungunya virus antigens, powder for suspension for injection, 5xE4 (± 0.5 log) TCID50/dose physiological saline solution: sterile physiological saline solution 0.9% used as placebo
- Treatment Group B/D; Priorix®: Participants received i.m. vaccinations with placebo on study day 0, Priorix® on day 28 and one boosting dose with Priorix® on day 196. Priorix®: lyophilized mixed preparation containing the attenuated Schwarz measles virus strain, the RIT 4385 strain of mumps virus (derived from the Jeryl Lynn strain) and the Wistar RA 27/3 rubella virus strain. Powder and solvent for suspension for injection physiological saline solution: sterile physiological saline solution 0.9% used as placebo
- Treatment Group C; MV-CHIK High: Participants received i.m. vaccinations with MV-CHIK high dose (5xE5 (± 0.5 log) TCID50 per 0.3 mL) on study day 0 and 28, placebo on day 196. MV-CHIK high dose: recombinant measles virus vaccine expressing Chikungunya virus antigens, powder for suspension for injection; 5xE5 (± 0.5 log) TCID50/dose physiological saline solution: sterile physiological saline solution 0.9% used as placebo
- Treatment Group D; MV-CHIK High: Participants received i.m. vaccinations with placebo on study day 0, MV-CHIK high dose (5xE5 (± 0.5 log) TCID50 per 0.3 mL) on study day 28 and MV-CHIK boosting dose on day 196. MV-CHIK high dose: recombinant measles virus vaccine expressing Chikungunya virus antigens, powder for suspension for injection; 5xE5 (± 0.5 log) TCID50/dose physiological saline solution: sterile physiological saline solution 0.9% used as placebo
- Measles Booster Group 1: Participants received i.m. vaccinations with Priorix® on study day -28, MV-CHIK on day 0 and 28 and placebo on day 168 and 196. MV-CHIK low dose: recombinant measles virus vaccine expressing Chikungunya virus antigens, powder for suspension for injection, 5xE4 (± 0.5 log) TCID50/dose Priorix®: lyophilized mixed preparation containing the attenuated Schwarz measles virus strain, the RIT 4385 strain of mumps virus (derived from the Jeryl Lynn strain) and the Wistar RA 27/3 rubella virus strain. Powder and solvent for suspension for injection physiological saline solution: sterile physiological saline solution 0.9% used as placebo
- Measles Booster Group 2: Participants received i.m. vaccinations with Priorix® on study day -28, placebo on day 0 and 28 and MV-CHIK on day 168 and 196. MV-CHIK low dose: recombinant measles virus vaccine expressing Chikungunya virus antigens, powder for suspension for injection, 5xE4 (± 0.5 log) TCID50/dose Priorix®: lyophilized mixed preparation containing the attenuated Schwarz measles virus strain, the RIT 4385 strain of mumps virus (derived from the Jeryl Lynn strain) and the Wistar RA 27/3 rubella virus strain. Powder and solvent for suspension for injection physiological saline solution: sterile physiological saline solution 0.9% used as placebo
Period: Overall Study
Arm/Group | Treatment Group A; MV-CHIK Low | Treatment Group A/C; Priorix® | Treatment Group B; MV-CHIK Low | Treatment Group B/D; Priorix® | Treatment Group C; MV-CHIK High | Treatment Group D; MV-CHIK High | Measles Booster Group 1 | Measles Booster Group 2
Started | 51 | 18 | 47 | 16 | 47 | 50 | 18 | 16
Completed | 47 | 15 | 46 | 16 | 47 | 45 | 17 | 16
Not Completed | 4 | 3 | 1 | 0 | 0 | 5 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 3 | 1 | 1 | 0 | 0 | 3 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Population as well as the Modified Intent-to-treat (mITT) population included all randomized subjects who received at least one vaccination and included 263 participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group A; MV-CHIK Low | Treatment Group A/C; Priorix® | Treatment Group B; MV-CHIK Low | Treatment Group B/D; Priorix® | Treatment Group C; MV-CHIK High | Treatment Group D; MV-CHIK High | Measles Booster Group 1 | Measles Booster Group 2 | Total
Number analyzed (Participants) | 51 | 18 | 47 | 16 | 47 | 50 | 18 | 16 | 263
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Demography and baseline characteristics include 263 participants of the mITT population
  years | 31.4 (10.13) | 32.2 (10.01) | 32.7 (10.53) | 33.6 (11.56) | 35.1 (12.32) | 31.2 (9.93) | 31.1 (10.41) | 32.6 (10.28) | 32.5 (10.65)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Demography and baseline characterisitcs of mITT Population including 263 subjects.
  Participants
    Female | 27 | 10 | 29 | 7 | 24 | 27 | 11 | 5 | 140
    Male | 24 | 8 | 18 | 9 | 23 | 23 | 7 | 11 | 123
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Demography and baseline characteristics including mITT Population of 263 participants
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
    White | 50 | 17 | 47 | 16 | 45 | 49 | 17 | 16 | 257
    More than one race | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Functional Anti-chikungunya Antibody Titers on Day 56 (28 Days Post Immunisation) Confirmed by Plaque Reduction Neutralization Test (PRNT50)
Description: Immunogenicity on day 56 confirmed by the presence of functional anti-chikungunya antibodies as determined by the plaque reduction neutralization test (PRNT50). This means immunogenicity 28 days after primary immunization regime, comprising one or two vaccinations.
Time Frame: Study day 56 (28 days after one or two vaccinations depending on treatment group).
Population: The Per-Protocol (PP) population was defined as the mITT population minus subjects with at least one major protocol deviation
Measure: Geometric Mean (Standard Deviation); unit: Titer
Arm/Group | Treatment Group A; MV-CHIK Low | Treatment Group A/C; Priorix® | Treatment Group B; MV-CHIK Low | Treatment Group B/D; Priorix® | Treatment Group C; MV-CHIK High | Treatment Group D; MV-CHIK High | Measles Booster Group 1 | Measles Booster Group 2
Number analyzed (Participants) | 49 | 16 | 44 | 2 | 47 | 44 | 16 | 15
Titer | 50.2 (127.69) | 5.0 (0.00) | 12.9 (100.47) | 5.0 (0.00) | 174.8 (436.11) | 33.6 (59.38) | 80.0 (233.80) | 5.0 (0.00)
Statistical Analysis 1: Comparison: Treatment Group A; MV-CHIK Low vs Treatment Group B; MV-CHIK Low; Test type: Superiority; p < 0.0001, ANOVA — Pairwise comparisons were adjusted for multiple tests according to Tukey-Kramer. The threshold for significance was 0.05; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 3.9, 95% CI 2-sided [2.0 to 7.7]
Statistical Analysis 2: Comparison: Treatment Group A; MV-CHIK Low vs Treatment Group C; MV-CHIK High; Test type: Superiority; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 0.3, 95% CI 2-sided [0.1 to 0.6]
Statistical Analysis 3: Comparison: Treatment Group A; MV-CHIK Low vs Treatment Group D; MV-CHIK High; Test type: Superiority; p = 0.6334, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 1.5, 95% CI 2-sided [0.8 to 3.0]
Statistical Analysis 4: Comparison: Treatment Group A; MV-CHIK Low vs Measles Booster Group 1; Test type: Superiority; p = 0.8065, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 0.6, 95% CI 2-sided [0.2 to 1.6]
Statistical Analysis 5: Comparison: Treatment Group A; MV-CHIK Low vs Measles Booster Group 2; Test type: Superiority; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 10.0, 95% CI 2-sided [3.8 to 26.6]
Statistical Analysis 6: Comparison: Treatment Group A; MV-CHIK Low vs Treatment Group A/C; Priorix®; Test type: Superiority; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 0.1, 95% CI 2-sided [0.0 to 0.3]
Statistical Analysis 7: Comparison: Treatment Group A; MV-CHIK Low vs Treatment Group B/D; Priorix®; Test type: Superiority; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 0.1, 95% CI 2-sided [0.0 to 0.3]
Statistical Analysis 8: Comparison: Treatment Group B; MV-CHIK Low vs Treatment Group C; MV-CHIK High; Test type: Superiority; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 0.1, 95% CI 2-sided [0.0 to 0.1]
Statistical Analysis 9: Comparison: Treatment Group B; MV-CHIK Low vs Treatment Group D; MV-CHIK High; Test type: Superiority; p = 0.0011, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 0.4, 95% CI 2-sided [0.2 to 0.8]
Statistical Analysis 10: Comparison: Treatment Group B; MV-CHIK Low vs Measles Booster Group 1; Test type: Superiority; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 0.2, 95% CI 2-sided [0.1 to 0.4]
Statistical Analysis 11: Comparison: Treatment Group B; MV-CHIK Low vs Measles Booster Group 2; Test type: Superiority; p = 0.0718, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 2.6, 95% CI 2-sided [1.0 to 6.9]
Statistical Analysis 12: Comparison: Treatment Group A/C; Priorix® vs Treatment Group B; MV-CHIK Low; Test type: Superiority; p = 0.0593, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 0.4, 95% CI 2-sided [0.1 to 1.0]
Statistical Analysis 13: Comparison: Treatment Group B; MV-CHIK Low vs Treatment Group B/D; Priorix®; Test type: Superiority; p = 0.0593, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of variance was conducted with treatment group as a fixed factor; Gemetric mean ratio = 0.4, 95% CI 2-sided [0.1 to 1.0]
Statistical Analysis 14: Comparison: Treatment Group C; MV-CHIK High vs Treatment Group D; MV-CHIK High; Test type: Superiority; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 5.2, 95% CI 2-sided [2.6 to 10.4]
Statistical Analysis 15: Comparison: Treatment Group C; MV-CHIK High vs Measles Booster Group 1; Test type: Superiority; p = 0.2005, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 2.2, 95% CI 2-sided [0.8 to 5.7]
Statistical Analysis 16: Comparison: Treatment Group C; MV-CHIK High vs Measles Booster Group 2; Test type: Superiority; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 35.0, 95% CI 2-sided [13.1 to 93.1]
Statistical Analysis 17: Comparison: Treatment Group A/C; Priorix® vs Treatment Group C; MV-CHIK High; Test type: Superiority; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 0.0, 95% CI 2-sided [0.0 to 0.1]
Statistical Analysis 18: Comparison: Treatment Group B/D; Priorix® vs Treatment Group C; MV-CHIK High; Test type: Superiority; p < 0.0001, ANOVA; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 0.0, 0.0% CI 2-sided [0.0 to 0.1]
Statistical Analysis 19: Comparison: Treatment Group D; MV-CHIK High vs Measles Booster Group 1; Test type: Superiority; p = 0.1138, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 0.4, 95% CI 2-sided [0.2 to 1.1]
Statistical Analysis 20: Comparison: Treatment Group D; MV-CHIK High vs Measles Booster Group 2; Test type: Superiority; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 6.7, 95% CI 2-sided [2.5 to 18.1]
Statistical Analysis 21: Comparison: Treatment Group A/C; Priorix® vs Treatment Group D; MV-CHIK High; Test type: Superiority; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 0.1, 95% CI 2-sided [0.1 to 0.4]
Statistical Analysis 22: Comparison: Treatment Group B/D; Priorix® vs Treatment Group D; MV-CHIK High; Test type: Superiority; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 0.1, 95% CI 2-sided [0.1 to 0.4]
Statistical Analysis 23: Comparison: Measles Booster Group 1 vs Measles Booster Group 2; Test type: Superiority; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 16.0, 95% CI 2-sided [4.9 to 52.4]
Statistical Analysis 24: Comparison: Treatment Group A/C; Priorix® vs Measles Booster Group 1; Test type: Superiority; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 0.1, 95% CI 2-sided [0.0 to 0.2]
Statistical Analysis 25: Comparison: Treatment Group B/D; Priorix® vs Measles Booster Group 1; Test type: Superiority; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 0.1, 95% CI 2-sided [0.0 to 0.2]
Statistical Analysis 26: Comparison: Treatment Group A/C; Priorix® vs Measles Booster Group 2; Test type: Superiority; p = 1.0000, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 1.0, 95% CI 2-sided [0.3 to 3.3]
Statistical Analysis 27: Comparison: Treatment Group B/D; Priorix® vs Measles Booster Group 2; Test type: Superiority; p = 1.0000, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 1.0, 95% CI 2-sided [0.3 to 3.3]
Statistical Analysis 28: Comparison: Treatment Group A/C; Priorix® vs Treatment Group B/D; Priorix®; Test type: Superiority; p = 1.0000, ANOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of variance was conducted with treatment group as a fixed factor; Geometric mean ratio = 1.0, 95% CI 2-sided [0.3 to 3.2]

2. Secondary Outcome: Functional Anti-Chikungunya Antibody Titers on Days 0, 28, 196 and 224 (M1/M2 Groups Day 168) Confirmed by Plaque Reduction Neutralization Test (PRNT50)
Description: Evaluation of immunogenicity on day 0, 28, 196 and 224; additionally for group M1 and M2 on day 168 as confirmed by the presence of functional anti-chikungunya antibodies, determined by the plaque reduction neutralization test (PRNT50).
Time Frame: Baseline until study day 224
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: Titer
Groups:
- Treatment Group B; MV-CHIK Low: Participants received i.m. vaccinations with placebo on study day 0. MV-CHIK low dose (5xE4 (± 0.5 log) TCID50 per 0.3 mL) on day 28 and MV-CHIK boosting dose on day 196. MV-CHIK low dose: recombinant measles virus vaccine expressing Chikungunya virus antigens, powder for suspension for injection, 5xE4 (± 0.5 log) TCID50/dose physiological saline solution: sterile physiological saline solution 0.9% used as placebo
Arm/Group | Treatment Group A; MV-CHIK Low | Treatment Group A/C; Priorix® | Treatment Group B; MV-CHIK Low | Treatment Group B/D; Priorix® | Treatment Group C; MV-CHIK High | Treatment Group D; MV-CHIK High | Measles Booster Group 1 | Measles Booster Group 2
Number analyzed (Participants) | 49 | 16 | 44 | 16 | 47 | 44 | 16 | 15
Titer
  Visit 1 /day 0 | 5.1 (0.71) | 5.0 (0.00) | 5.3 (3.16) | 5.0 (0.00) | 5.0 (0.00) | 5.0 (0.00) | 5.0 (0.00) | 5.0 (0.00)
  Visit 2 /day 28 | 11.2 (63.40) | 5.0 (0.00) | 5.5 (3.82) | 5.0 (0.00) | 25.7 (52.22) | 5.1 (0.75) | 13.5 (40.52) | 5.0 (0.00)
  Visit 4 /day 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 15
  Visit 4 /day 168 |  |  |  |  |  |  | 28.9 (52.25) | 5.0 (0.00)
  Visit 5 /day 196: number analyzed (Participants) | 46 | 15 | 44 | 16 | 47 | 43 | 15 | 15
  Visit 5 /day 196 | 13.5 (33.46) | 5.0 (0.00) | 6.4 (8.29) | 5.00 (0.00) | 38.8 (70.59) | 16.5 (81.75) | 24.1 (106.25) | 11.5 (26.04)
  Visit 6 /day 224 | 14.6 (37.87) | 5.0 (0.00) | 70.5 (174.57) | 5.0 (0.00) | 41.8 (105.55) | 609.8 (949.70) | 18.3 (87.50) | 66.5 (172.62)

3. Secondary Outcome: Measurement of Anti-measles Antibody Titer by Enzyme Linked Immunosorbent Assay
Description: Determination of anti-measles antibodies on day 0, 28, and 56; additionally for group M1 and M2 on day -28 by enzyme linked immunosorbent assay (ELISA).
Time Frame: Baseline until study day 56
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: Titer
Arm/Group | Treatment Group A; MV-CHIK Low | Treatment Group A/C; Priorix® | Treatment Group B; MV-CHIK Low | Treatment Group B/D; Priorix® | Treatment Group C; MV-CHIK High | Treatment Group D; MV-CHIK High | Measles Booster Group 1 | Measles Booster Group 2
Number analyzed (Participants) | 49 | 16 | 44 | 16 | 47 | 44 | 16 | 15
Titer
  Visit 0 / day -28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 15
  Visit 0 / day -28 |  |  |  |  |  |  | 542.6 (1118.52) | 304.5 (343.53)
  Visit 1 / day 0 | 456.2 (1398.54) | 693.9 (1307.42) | 398.1 (1267.55) | 390.4 (1106.86) | 495.0 (1181.36) | 401.8 (1073.54) | 785.6 (1149.47) | 645.9 (850.56)
  Visit 2 / day 28 | 1509.4 (1360.83) | 1200.6 (1129.77) | 396.9 (1183.04) | 447.5 (1139.37) | 2343.9 (1357.29) | 492.1 (1227.24) | 1761.5 (1578.85) | 561.2 (385.36)
  Visit 3 / day 56 | 1651.8 (1384.39) | 1129.4 (1168.63) | 1255.0 (1279.28) | 673.8 (917.52) | 2750.5 (1284.23) | 2435.2 (1461.78) | 1825.2 (1459.93) | 521.4 (455.37)

4. Secondary Outcome: Number of Participants With Solicited Local and Systemic Adverse Events
Description: Evaluation of solicited local and systemic adverse events as recorded in the subjects' diaries for 7 days after each vaccination. As per the protocol, adverse events were analyzed per treatment group but were not assessed with respect to individual vaccinations.
Time Frame: Solicited adverse events were recorded for 7 days after each vaccination
Population: All safety analyses were based on the Safety Population, which included all subjects who received at least one vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group A; MV-CHIK Low | Treatment Group A/C; Priorix® | Treatment Group B; MV-CHIK Low | Treatment Group B/D; Priorix® | Treatment Group C; MV-CHIK High | Treatment Group D; MV-CHIK High | Measles Booster Group 1 | Measles Booster Group 2
Number analyzed (Participants) | 51 | 18 | 47 | 16 | 47 | 50 | 18 | 16
Participants | 35 | 14 | 32 | 10 | 37 | 41 | 13 | 10

5. Secondary Outcome: Number of Participants Who Experienced Treatment Emergent Adverse Events
Description: Evaluation of all treatment emergent adverse events (TEAEs) occurred throughout the clinical study. Clinically relevant abnormal safety laboratory values were recorded as TEAEs. As per the protocol, adverse events were analyzed per treatment group but were not assessed with respect to individual vaccinations.
Time Frame: First vaccination until study day 224
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group A; MV-CHIK Low | Treatment Group A/C; Priorix® | Treatment Group B; MV-CHIK Low | Treatment Group B/D; Priorix® | Treatment Group C; MV-CHIK High | Treatment Group D; MV-CHIK High | Measles Booster Group 1 | Measles Booster Group 2
Number analyzed (Participants) | 51 | 18 | 47 | 16 | 47 | 50 | 18 | 16
Participants
  TEAEs | 29 | 10 | 27 | 7 | 22 | 18 | 11 | 9
  Serious TEAEs | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 0
  Severe TEAEs | 1 | 1 | 2 | 0 | 0 | 2 | 1 | 1
  Related TEAEs | 8 | 2 | 11 | 1 | 4 | 10 | 4 | 5
  Medically attended TEAEs | 12 | 3 | 15 | 1 | 9 | 8 | 4 | 3
  TEAEs where an action was taken | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
  TEAEs of special interest | 2 | 0 | 2 | 0 | 0 | 1 | 2 | 0

6. Secondary Outcome: Number of Participants With Shedding of Live Recombinant Virus in Urine Until Day 196
Description: Shedding was observed in a subset of subjects at one Austrian study site, by qualitative determination of live recombinant measles virus in urine by polymerase chain reaction (PCR).
Time Frame: Baseline until study day 196; assessed on days 0, 7, 10, 14, 28 and 196
Population: As subjects of the measles booster groups M1 and M2 received a measles vaccination prior to the modified MV-CHIK vaccine, these groups had to be excluded from measles shedding analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group A; MV-CHIK Low | Treatment Group A/C; Priorix® | Treatment Group B; MV-CHIK Low | Treatment Group B/D; Priorix® | Treatment Group C; MV-CHIK High | Treatment Group D; MV-CHIK High | Measles Booster Group 1 | Measles Booster Group 2
Number analyzed (Participants) | 8 | 4 | 4 | 2 | 8 | 5 | 0 | 0
Participants
  Visit 1 /day 0: number analyzed (Participants) | 7 | 4 | 3 | 2 | 8 | 4 | 0 | 0
  Visit 1 /day 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  day 7: number analyzed (Participants) | 8 | 3 | 3 | 2 | 8 | 5 | 0 | 0
  day 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  day 10: number analyzed (Participants) | 8 | 4 | 4 | 2 | 6 | 3 | 0 | 0
  day 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  day 14: number analyzed (Participants) | 8 | 3 | 4 | 1 | 7 | 5 | 0 | 0
  day 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Visit 2 /day 28 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Visit 5 /day 196: number analyzed (Participants) | 8 | 3 | 4 | 2 | 8 | 5 | 0 | 0
  Visit 5 /day 196 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Shedding of Live Recombinant Virus in Saliva Until Day 196
Description: Shedding was observed in a subset of subjects at one Austrian study site, by qualitative determination of live recombinant measles virus in saliva by polymerase chain reaction (PCR).
Time Frame: Baseline until study day 196; assessed on days 0, 7, 10, 14, 28 and 196
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group A; MV-CHIK Low | Treatment Group A/C; Priorix® | Treatment Group B; MV-CHIK Low | Treatment Group B/D; Priorix® | Treatment Group C; MV-CHIK High | Treatment Group D; MV-CHIK High | Measles Booster Group 1 | Measles Booster Group 2
Number analyzed (Participants) | 8 | 4 | 4 | 2 | 8 | 5 | 0 | 0
Participants
  Visit 1/Day 0: number analyzed (Participants) | 8 | 4 | 3 | 2 | 8 | 5 | 0 | 0
  Visit 1/Day 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 7: number analyzed (Participants) | 8 | 3 | 3 | 2 | 8 | 5 | 0 | 0
  Day 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 10: number analyzed (Participants) | 8 | 4 | 4 | 2 | 7 | 3 | 0 | 0
  Day 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 14: number analyzed (Participants) | 8 | 3 | 4 | 1 | 7 | 5 | 0 | 0
  Day 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Visit 2/Day 28 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Visit 5/Day 196: number analyzed (Participants) | 8 | 3 | 4 | 2 | 8 | 5 | 0 | 0
  Visit 5/Day 196 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Chikungunya Virus Specific T Cell Responses
Description: Peripheral blood mononuclear cells (PBMCs) were isolated from whole blood to determine functional IL-2-producing T cells on day 0, 28, 56 and 224 in a subset of subjects. ELISpots were performed using peptides covering the CHIK proteins E1, E2 and C for re-stimulation, thereby producing three values per sample representing the number of spots per 1 x 10^6 PBMCs. If one or more of the three values was greater than 50, the sample was considered positive and the highest of the three values was used in the analysis. If all three values were below 50, the sample was considered negative and a value of 0.0 was used for analysis.
Time Frame: Baseline until study day 224
Population: A subset of the mITT Population was analyzed for T-cell Response.
Measure: Mean (Standard Deviation); unit: Titer
Arm/Group | Treatment Group A; MV-CHIK Low | Treatment Group A/C; Priorix® | Treatment Group B; MV-CHIK Low | Treatment Group B/D; Priorix® | Treatment Group C; MV-CHIK High | Treatment Group D; MV-CHIK High | Measles Booster Group 1 | Measles Booster Group 2
Number analyzed (Participants) | 51 | 18 | 47 | 16 | 47 | 50 | 18 | 16
Titer
  Visit 1 /day 0: number analyzed (Participants) | 11 | 5 | 11 | 4 | 12 | 11 | 2 | 0
  Visit 1 /day 0 | 0.0 (0.00) | 0.0 (0.00) | 12.1 (40.10) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) |
  Visit 2 /day 28: number analyzed (Participants) | 15 | 5 | 0 | 0 | 14 | 0 | 0 | 0
  Visit 2 /day 28 | 41.5 (128.71) | 0.0 (0.00) |  |  | 10.5 (39.29) |  |  |
  Visit 3 /day 56: number analyzed (Participants) | 14 | 5 | 12 | 5 | 14 | 11 | 5 | 4
  Visit 3 /day 56 | 46.5 (63.54) | 0.0 (0.00) | 36.7 (68.41) | 25.2 (56.35) | 53.4 (74.38) | 6.5 (21.41) | 47.0 (51.55) | 0.0 (0.00)
  Visit 6 /day 224: number analyzed (Participants) | 15 | 5 | 12 | 5 | 14 | 10 | 5 | 4
  Visit 6 /day 224 | 28.3 (48.92) | 0.0 (0.00) | 71.8 (133.03) | 13.2 (29.52) | 11.6 (23.06) | 30.1 (61.48) | 0.0 (0.00) | 0.0 (0.00)

9. Secondary Outcome: Immunogenicity Confirmed by the Presence of Humoral Anti-chikungunya Antibodies, Determined by Enzyme Linked Immunosorbent Assay (ELISA)
Description: Evaluation of immunogenicity mediated by serum IgG antibodies against Chikungunya on days 0, 28, 196 and 224; additionally for group M1 and M2 on day 168, determined by enzyme linked immunosorbent assay (ELISA).
Time Frame: Baseline until study day 224; assessed on days 0, 28, 168, 196 and 224
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: Titer
Arm/Group | Treatment Group A; MV-CHIK Low | Treatment Group A/C; Priorix® | Treatment Group B; MV-CHIK Low | Treatment Group B/D; Priorix® | Treatment Group C; MV-CHIK High | Treatment Group D; MV-CHIK High | Measles Booster Group 1 | Measles Booster Group 2
Number analyzed (Participants) | 49 | 16 | 44 | 16 | 47 | 44 | 16 | 15
Titer
  Visit 1 /day 0 | 2.1 (1.94) | 3.6 (3.64) | 2.3 (1.68) | 1.7 (1.05) | 2.3 (2.75) | 2.2 (1.53) | 2.4 (2.69) | 2.2 (2.25)
  Visit 2 /day 28 | 3.2 (6.57) | 3.4 (3.13) | 2.2 (1.81) | 2.0 (2.75) | 6.2 (4.65) | 2.5 (1.74) | 4.3 (9.48) | 2.0 (2.37)
  Visit 3 /day 56 | 13.6 (31.84) | 3.4 (4.06) | 3.4 (6.26) | 1.7 (1.63) | 74.4 (41.45) | 6.6 (18.68) | 28.0 (47.51) | 2.3 (2.10)
  Visit 4 /day 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 15
  Visit 4 /day 168 |  |  |  |  |  |  | 9.5 (29.82) | 1.8 (2.28)
  Visit 5 /day 196: number analyzed (Participants) | 46 | 15 | 44 | 16 | 47 | 43 | 16 | 15
  Visit 5 /day 196 | 5.6 (16.04) | 3.3 (4.02) | 3.0 (3.11) | 1.9 (2.06) | 15.2 (25.08) | 5.6 (21.33) | 8.9 (24.13) | 3.6 (5.48)
  Visit 6 /day 224: number analyzed (Participants) | 46 | 15 | 44 | 16 | 47 | 43 | 16 | 15
  Visit 6 /day 224 | 4.6 (9.46) | 3.1 (4.66) | 25.4 (52.43) | 1.7 (1.82) | 13.1 (24.24) | 130.8 (43.94) | 7.3 (28.56) | 20.4 (43.19)

10. Secondary Outcome: Functional Anti-chikungunya Antibody Titers on Day 56 (28 Days Post Immunization) by Baseline Measles Titer
Description: To determine the potential impact of pre-existing antibodies against measles on MV-CHIK immunogenicity, participants from treatment Groups A to D were divided into quartiles according to serum IgG concentrations against measles virus on Day 0. Functional anti-chikungunya antibodies as determined by PRNT50 were compared between groups.
Time Frame: Study day 56 (28 days after one or two vaccinations depending on treatment group)
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: Titer
Groups:
- Baseline Measles Titer Percentile 0 to 25%; Baseline Measles Titer Percentile 25 to 50%; Baseline Measles Titer Percentile 50 to 75%; Baseline Measles Titer Percentile 75 to 100%: Participants in Treatment Groups A, B, C, and D categorized according to baseline measles titer value.
Arm/Group | Baseline Measles Titer Percentile 0 to 25% | Baseline Measles Titer Percentile 25 to 50% | Baseline Measles Titer Percentile 50 to 75% | Baseline Measles Titer Percentile 75 to 100%
Number analyzed (Participants) | 45 | 48 | 45 | 46
Titer | 155.1 (532.68) | 177.0 (897.74) | 117.6 (346.86) | 100.8 (535.78)
Statistical Analysis 1: Comparison: Baseline Measles Titer Percentile 0 to 25% vs Baseline Measles Titer Percentile 25 to 50%; Test type: Superiority; p = 0.9775, ANOVA; Analysis of variance was performed with baseline measles titer group as a fixed factor; Geometric mean ratio = 0.9, 95% CI 2-sided [0.4 to 2.0]
Statistical Analysis 2: Comparison: Baseline Measles Titer Percentile 0 to 25% vs Baseline Measles Titer Percentile 50 to 75%; Test type: Superiority; p = 0.8366, ANOVA; Analysis of variance was performed with baseline measles titer group as a fixed factor; Geometric mean ratio = 1.3, 95% CI 2-sided [0.6 to 3.1]
Statistical Analysis 3: Comparison: Baseline Measles Titer Percentile 0 to 25% vs Baseline Measles Titer Percentile 75 to 100%; Test type: Superiority; p = 0.5625, ANOVA; Analysis of variance was performed with baseline measles titer group as a fixed factor; Geometric mean ratio = 1.5, 95% CI 2-sided [0.7 to 3.6]
Statistical Analysis 4: Comparison: Baseline Measles Titer Percentile 25 to 50% vs Baseline Measles Titer Percentile 50 to 75%; Test type: Superiority; p = 0.5924, ANOVA; Analysis of variance was performed with baseline measles titer group as a fixed factor; Geometric mean ratio = 1.5, 95% CI 2-sided [0.6 to 3.5]
Statistical Analysis 5: Comparison: Baseline Measles Titer Percentile 25 to 50% vs Baseline Measles Titer Percentile 75 to 100%; Test type: Superiority; p = 0.3122, ANOVA; Analysis of variance was performed with baseline measles titer group as a fixed factor; Geometric mean ratio = 1.8, 95% CI 2-sided [0.8 to 4.1]
Statistical Analysis 6: Comparison: Baseline Measles Titer Percentile 50 to 75% vs Baseline Measles Titer Percentile 75 to 100%; Test type: Superiority; p = 0.9665, ANOVA; Analysis of variance was performed with baseline measles titer group as a fixed factor; Geometric mean ratio = 1.2, 95% CI 2-sided [0.5 to 2.8]

ADVERSE EVENTS:
Time Frame: 32 - 36 weeks Adverse events were collected in the period after the first vaccination until the last on site study visit.
Description: Local and systemic solicited adverse events were collected via subject diary, for 7 days after each vaccination. As per the protocol, adverse events were analyzed per treatment group but were not assessed with respect to individual vaccinations.
Arm/Group | Treatment Group A; MV-CHIK Low | Treatment Group A/C; Priorix® | Treatment Group B; MV-CHIK Low | Treatment Group B/D; Priorix® | Treatment Group C; MV-CHIK High | Treatment Group D; MV-CHIK High | Measles Booster Group 1 | Measles Booster Group 2
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/18 | 0/47 | 0/16 | 0/47 | 0/50 | 0/18 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/51 | 1/18 | 2/47 | 1/16 | 0/47 | 1/50 | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 40/51 | 14/18 | 36/47 | 11/16 | 38/47 | 41/50 | 15/18 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group A; MV-CHIK Low (N=51) | Treatment Group A/C; Priorix® (N=18) | Treatment Group B; MV-CHIK Low (N=47) | Treatment Group B/D; Priorix® (N=16) | Treatment Group C; MV-CHIK High (N=47) | Treatment Group D; MV-CHIK High (N=50) | Measles Booster Group 1 (N=18) | Measles Booster Group 2 (N=16)
umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 — rupture cruciate ligament left knee
abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 — suspected abortion
papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 — papillary thyroid carcinoma
laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 — larynx carcinoma
type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 — diabetes mellitus type 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group A; MV-CHIK Low (N=51) | Treatment Group A/C; Priorix® (N=18) | Treatment Group B; MV-CHIK Low (N=47) | Treatment Group B/D; Priorix® (N=16) | Treatment Group C; MV-CHIK High (N=47) | Treatment Group D; MV-CHIK High (N=50) | Measles Booster Group 1 (N=18) | Measles Booster Group 2 (N=16)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 13 (17) | 4 (4) | 9 (12) | 1 (1) | 9 (12) | 8 (16) | 2 (2) | 4 (7)
Fatigue (General disorders) | 10 (15) | 5 (9) | 9 (20) | 3 (5) | 13 (19) | 14 (25) | 5 (10) | 4 (9)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 1 (3) | 0 (0) | 1 (2) | 2 (8) | 2 (4) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 4 (5) | 1 (1) | 2 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 20 (36) | 10 (19) | 16 (32) | 6 (13) | 14 (30) | 17 (47) | 9 (18) | 8 (19)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (8) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (12) | 5 (8) | 6 (9) | 2 (2) | 5 (7) | 13 (22) | 4 (8) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appetite disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 7 (7) | 2 (2) | 4 (4) | 2 (3) | 4 (5) | 4 (5) | 2 (5) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 2 (3) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 3 (4) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 6 (8) | 2 (3) | 5 (6) | 2 (2) | 10 (18) | 9 (11) | 2 (4) | 2 (2)
Injection site induration (General disorders) | 5 (7) | 0 (0) | 6 (6) | 0 (0) | 8 (12) | 15 (24) | 2 (2) | 1 (1)
Injection site oedema (General disorders) | 4 (8) | 0 (0) | 2 (2) | 0 (0) | 3 (4) | 4 (6) | 1 (2) | 1 (1)
Injection site pain (General disorders) | 24 (51) | 6 (12) | 21 (37) | 5 (7) | 30 (71) | 39 (119) | 8 (29) | 7 (18)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 3 (4) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (10) | 4 (7) | 2 (3) | 2 (2) | 2 (2) | 6 (7) | 2 (2) | 1 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (9) | 3 (3) | 5 (7) | 2 (2) | 2 (2) | 7 (11) | 2 (3) | 3 (3)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertabral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3) | 5 (7) | 2 (2) | 4 (4) | 11 (19) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT02861586/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/86/NCT02861586/SAP_001.pdf